CLINICAL TRIAL: NCT05443269
Title: Impact of Jump Start Nutrition Program on Weight Loss and Associated Measures of Health in Overweight and Obese Men and Women
Brief Title: Impact of Jump Start Nutrition Program on Weight Loss and Associated Measures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Memphis (Other)
Collaborators: USANA Health Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PRO-FY2022-183
Record Dates: First submitted 2022-06-29; First posted 2022-07-05 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Weight Loss
Keywords: Jump Start; USANA
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Jump Start Program (Experimental): The intervention consists of following the Jump Start plan for 7 days
  Interventions: Dietary Supplement: Jump Start Nutritional Program

INTERVENTIONS:
Dietary Supplement: Jump Start Nutritional Program — Nutri-meal Active meal replacement shake and Metabolism pill at breakfast, lunch, and dinner, morning and evening Health Pak (multivitamin), 1 probiotic stick, and 300 calories fruits and vegetables daily

SUMMARY:
The purpose of the proposed study is to evaluate the impact of the Jump Start program to facilitate weight loss in a sample of overweight and obese men and women. The study will not only evaluate weight loss and changes in body-shape but will also assess the type of weight lost (fat vs. lean mass) and other health measures affected by obesity including lipids, glucose, insulin, resting heart rate and blood pressure, and perceived wellness. This study will contribute to the general weight loss literature by providing evidence for or against the use of a meal replacement centered one-week weight loss program to yield weight loss and other health-specific benefits. The hypothesis is that the Jump Start program will result in an average 3-5 pound weight loss, as well as improvements in bloodborne markers of health, from day 1 to day 8.

ELIGIBILITY:
Inclusion Criteria:

* BMI of 28-39.9 kg/m2
* can fast >10 hours
* maintain existing exercise regiment during study

Exclusion Criteria:

* Weight greater than 500 lbs
* Type I or II diabetic
* liver disease
* tobacco user
* adversity to fiber or protein supplement
* taking weight loss dietary supplements or adhering to any weight loss plan in the month prior to and during participation in the study
* taking a multi-vitamin or pro-biotic, or if they were not recommended by a doctor, willing to stop for 4 weeks prior to the study.
* consumption of alcohol or caffeine within 24 hours of each testing visit
* strenuous exercise during the 24 hours period before each testing visit
* self-reported active infection or illness of any kind
* pregnant or lactating

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-02-14 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Body Composition | Day 8
  Changes in body composition as measured by dual-energy X-ray absorptiometry from baseline
Lipids Panel | Day 8
  Changes in lipids panel from baseline
Glucose | Day 8
  Changes in glucose from baseline
Insulin | Day 8
  Changes in insulin from baseline
Body Weight | Day 8
  Changes in body weight from baseline
Body Mass Index | Day 8
  Changes in body mass index from baseline
Resting Blood pressure | Day 8
  Changes in resting blood pressure from baseline
Resting Heart Rate | Day 8
  Changes in resting heart rate from baseline
Subjects' perceived wellness | Day 8
  Changes in subjects perceived wellness from baseline using a visual analog scale from 0 to 10 with 0 being very low and 10 being extremely high
Hip Circumference | Day 8
  Changes in hip circumference from baseline
Waist Circumference | Day 8
  Changes in waist circumference from baseline
Physical Appearance | Day 8
  Changes in physical appearance of trunk region from bottom of neck to knee region

SECONDARY OUTCOMES:
Diet | Day 8
  Changes in diet from before intervention determined using food logs

CONTACTS AND LOCATIONS:
Overall Officials: Jacquelyn Pence, PhD, Principal Investigator — Research Assistant Professor
Locations (1):
- Center for Nutraceutical and Dietary Supplement Research, Memphis, Tennessee, United States